CLINICAL TRIAL: NCT02336373
Title: SC Youth Treatment With Hydroxyurea Effects
Brief Title: Treatment of Hemoglobin SC Disease With Hydroxyurea
Acronym: SCYTHE
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: low enrollment
Sponsor: Baylor College of Medicine (Other)
Responsible Party: Principal Investigator, Vivien Sheehan, Assistant Professor, Baylor College of Medicine
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: H-35010 SCYTHE
Record Dates: First submitted 2015-01-08; First posted 2015-01-13 (Estimated); Results first posted 2020-09-09 (Actual); Last update posted 2020-09-09 (Actual); Status verified 2020-09

CONDITIONS: Hemoglobin SC Disease
Keywords: Hemoglobin SC disease; hydroxyurea; quality of life; viscosity; red cell density
MeSH Terms: conditions — Hemoglobin SC Disease | interventions — Hydroxyurea

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Hydroxurea (Experimental): Initiate hydroxyurea at 10 mg/kg daily and escalate hydroxyurea dose by 5 mg/kg/day every 8 weeks up to a maximum dose of 35 mg/kg/day if blood counts meet escalation criteria on at least 2 blood tests over eight weeks prior to dose increase.
  Interventions: Drug: hydroxyurea

INTERVENTIONS:
Drug: hydroxyurea — Treat symptomatic HbSC patients to MTD on hydroxyurea, and assess for clinical improvement using the PedsQL™ Sickle Cell Disease Module version 3.0 after 6 months at MTD, compared to entrance scores
  Other Names: Hydrea; Droxia

SUMMARY:
Sickle cell disease (SCD), specifically hemoglobin SC disease (HbSC), is a subtype of sickle cell disease with typically higher hemoglobin and milder or later disease complications. Sickle cell disease is a disorder in which red blood cells (RBCs) are abnormally shaped. This can result in painful episodes, serious infections, and damage to body organs. One medication used to treat sickle cell disease is hydroxyurea.

Hydroxyurea therapy offers significant benefits for infants, children, and adolescents with sickle cell anemia. These include a reduction in the frequency of pain crises and acute chest syndrome (inflammation of the lungs). Hydroxyurea has been given to many HbSC patients but HbSC patients were not included in the large clinical trials used to test hydroxyurea in SCD, so less is known about how HbSC patients respond to hydroxyurea.

The purpose of this research study is to see if hydroxyurea, a medication given to many children with the most common type of sickle cell, those who are homozygous for the sickle mutation (HbSS), helps children who have HbSC. The investigators will see if it helps by giving a questionaire when the medication is started, and then every two months at a clinic visit. The questionaire, called the Pediatric Quality of Life Inventory (PedsQL™) Sickle Cell Disease Module version 3.0, measures quality of life. The investigators will also see how hydroxyurea changes laboratory test numbers, and blood thickness.

DETAILED DESCRIPTION:
To be eligible to participate in this study, patients must have HbSC disease, have experienced a sickle cell disease related complication, or have a score of 80 or lower on the PedsQL™ Sickle Cell Disease Module version 3.0. This questionnaire will be offered to all patients with HbSC seen in our clinic that consent to this study. If the patient is sexually active, they will be offered birth control. If the patient chooses not to initiate effective birth control, they will be tested at their scheduled vist with a urine pregnancy test. If the patient becomes pregnant they will be removed from the study.

The maximum time patients will be on the study is 12 months after starting hydroxyurea therapy, with an option to participate in a 2 year observation study following the end of the study.

Patients will be assessed in the clinic every two months after starting treatment. Hydroxyurea will be started at 10 mg/kg/day, and increased by 5 mg/kg/day at eight week intervals if needed to reach a maximum tolerated dose (MTD). The most common side effect of the drug is a drop in infection fighting cells, or white blood cells, so the medication will be started at a low dose and the dose will be increased only if it is safe to do so.

Patients will be asked to allow the investigators to review information from their medical records at the start of the study, and throughout the study. If the patient would like to participate in the two year follow-up, their records will be reviewed during that period as well.

ELIGIBILITY:
Inclusion Criteria:

1. Diagnosis of HbSC disease
2. Score equal or lower than 80 on the PedsQL™ Sickle Cell Disease Module version 3.0
3. Have experienced a sickle cell disease related complication

Exclusion Criteria:

1. Failure to meet inclusion criteria.
2. Hydroxyurea usage in the last 3 months.
3. Chronic RBC transfusion therapy.
4. Packed red blood cell transfusion in the last 3 months (temporary exclusion).
5. Pregnancy, or refusal to use medically effective birth control if female and sexually active.

Ages: 5 Years to 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 32 (Actual)
Dates: Start 2014-12; Primary Completion 2017-02 (Actual); Study Completion 2017-03-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Vivien Sheehan, MD, Principal Investigator — Baylor College of Medicine
Locations (1):
- Texas Children's Hospital, Houston, Texas, United States

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Hydroxurea
Started | 32
Completed | 14
Not Completed | 18
Not completed — Protocol closed early | 4
Not completed — Physician Decision | 14

BASELINE CHARACTERISTICS:
Groups:
- Hydroxyurea: hydroxyurea (HU) at 10 mg/kg daily
Arm/Group | Hydroxyurea
Number analyzed (Participants) | 32
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 32
  Between 18 and 65 years | 0
  >=65 years | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 11 (3.5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 13
  Male | 19
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1
  Not Hispanic or Latino | 31
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 31
  White | 0
  More than one race | 1
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 32
PedsQLTM 3.0 SCD Module score [Mean (Standard Deviation); unit: units on a scale] — PedsQLTM 3.0 Sickle Cell Disease Module score
  units on a scale | 54.9 (20.4)

OUTCOME MEASURES:

1. Primary Outcome: Change in PedsQL SCDM
Description: Mean change in PedsQL™ Sickle Cell Disease Module version 3.0 score after achieving MTD compared with baseline.
  PedsQL™ Sickle Cell Disease Module version 3.0 scores are on a 100 point scale ranging from 0 to 100 with higher values indicating better quality of life.
  PedsQL: pediatric qulaity of life
Time Frame: 6 months
Population: Participants who achieved MTD of hydroxyureq per protocol with observed PEDSQL scores at 6-months and baseline (study entry).
Measure: Mean (Standard Deviation); unit: Score on PedsQL 3.0 SCD Module
Arm/Group | Hydroxurea
Number analyzed (Participants) | 6
Score on PedsQL 3.0 SCD Module | 5.7 (15.5)

2. Secondary Outcome: Change in HVR at 45s-1
Description: Change in hematocrit to viscosity ratio (HVR) at 45s-1 at follow-up versus baseline. This is a measure of oxygen carrying capacity, as a higher hematocrit with lower viscosity indicates ability to deliver oxygen without slowed blood flow due to high viscosity or blood thickness. Higher values are associated with improvement.
Time Frame: up to 7 months
Measure: Mean (Standard Deviation); unit: au
Groups:
- Hydroxyurea: Inititiate hydroxyurea and reach MTD
Arm/Group | Hydroxyurea
Number analyzed (Participants) | 6
au | 0.083 (0.72)

3. Secondary Outcome: Change in HVR at 225s-1
Description: Change in hematocrit viscosity ratio at 225s
Time Frame: up to 7 months
Measure: Mean (Standard Deviation); unit: au
Arm/Group | Hydroxyurea
Number analyzed (Participants) | 6
au | 0.11 (0.83)

4. Secondary Outcome: DRBC
Description: Change in percent dense red blood cells
Time Frame: up to 7 months
Measure: Mean (Standard Deviation); unit: percentage of dense red blood cells
Arm/Group | Hydroxyurea
Number analyzed (Participants) | 6
percentage of dense red blood cells | 1.93 (20.6)

5. Secondary Outcome: Change in HbF
Description: Change in fetal hemaglobin
Time Frame: up to 7 months
Measure: Mean (Standard Deviation); unit: percent
Arm/Group | Hydroxyurea
Number analyzed (Participants) | 6
percent | -0.47 (0.94)

6. Secondary Outcome: Change in MCV
Description: Change in mean corpuscular volume
Time Frame: up to 7 months
Measure: Mean (Standard Deviation); unit: fL
Arm/Group | Hydroxyurea
Number analyzed (Participants) | 6
fL | -6.2 (2.3)

7. Secondary Outcome: Change in MCHC
Description: Change in mean corpuscular hemoglobin concentration
Time Frame: up to 7 months
Measure: Mean (Standard Deviation); unit: percent
Arm/Group | Hydroxyurea
Number analyzed (Participants) | 6
percent | 0.33 (0.43)

8. Secondary Outcome: Change in Hb
Description: Change in hemoglobin
Time Frame: up to 7 months
Measure: Mean (Standard Deviation); unit: percent
Arm/Group | Hydroxyurea
Number analyzed (Participants) | 6
percent | -0.62 (0.59)

9. Secondary Outcome: Change in ARC
Description: Change in absolute reticulocyte count
Time Frame: up to 7 months
Measure: Mean (Standard Deviation); unit: 10^3 cells/uL
Arm/Group | Hydroxyurea
Number analyzed (Participants) | 6
10^3 cells/uL | 0.01 (0.025)

10. Secondary Outcome: Change in ANC
Description: Change in absolute neutrophil count
Time Frame: up to 7 months
Measure: Mean (Standard Deviation); unit: 10^3 cells/uL
Arm/Group | Hydroxyurea
Number analyzed (Participants) | 6
10^3 cells/uL | -0.24 (0.82)

11. Secondary Outcome: Change in LDH
Description: Change in lactate dehydrogenase
Time Frame: up to 7 months
Measure: Mean (Standard Deviation); unit: percent
Arm/Group | Hydroxyurea
Number analyzed (Participants) | 6
percent | -21.7 (52.48)

12. Secondary Outcome: Change in UB Levels
Description: Change in unconjugated bilirubin levels
Time Frame: up to 7 months
Measure: Mean (Standard Deviation); unit: percent
Arm/Group | Hydroxyurea
Number analyzed (Participants) | 5
percent | -0.1 (0.28)

ADVERSE EVENTS:
Time Frame: 1 year
Arm/Group | Hydroxurea
All-Cause Mortality (participants affected / at risk) | 0/32
Serious Adverse Events (participants affected / at risk) | 0/32
Other Adverse Events (participants affected / at risk) | 0/32

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2015-06-08): https://cdn.clinicaltrials.gov/large-docs/73/NCT02336373/Prot_SAP_000.pdf